CLINICAL TRIAL: NCT03427853
Title: A Randomized, Double-blind, Parallel-group, Placebo-controlled, Single-dose Escalation Phase I Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Immunogenicity of Denosumab Injection Administered Subcutaneously to Healthy Adults in China
Brief Title: A Study to Evaluate the Denosumab in Healthy Adults
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Luye Pharma Group Ltd. (Industry)
Collaborators: Shandong Boan Biotechnology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LY06006
Record Dates: First submitted 2018-01-31; First posted 2018-02-09 (Actual); Last update posted 2018-02-09 (Actual); Status verified 2018-02

CONDITIONS: Healthy Adults

STUDY DESIGN:
Intervention Model Description: randomized, double-blind, parallel-group, placebo-controlled, single-dose escalation
Who Masked: Participant, Investigator
Masking Description: double-blind,
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LY06006 (Experimental): LY06006 18mg, 60mg 120mg subcutaneous injection
  Interventions: Drug: LY06006
- Placebo (Placebo Comparator): Placebo subcutaneous injection
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: LY06006 — LY06006 18mg, 60mg, 120mg subcutaneous injection
  Arms: LY06006
Drug: Placebos — Placebo subcutaneous injection
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, parallel-group, placebo-controlled, single-dose escalation Phase I study to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics and immunogenicity of denosumab injection administered subcutaneously to healthy adults in China

DETAILED DESCRIPTION:
This is a randomized, double-blind, parallel-group, placebo-controlled, single-dose escalation Phase I study in healthy adults in China, conducted in one center.

The objectives are to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics and immunogenicity of denosumab injection (code name:LY06006).

Subjects would be sequentially enrolled in one of three cohorts. Eight subjects in the first cohort would receive a single 18 mg subcutaneous injection of LY06006. If the safety and tolerability were confirmed at Day 56, the other 16 subjects would be enrolled in the second cohort to receive a single 60 mg subcutaneous injection of LY06006. If the safety and tolerability were confirmed at Day 56 in 60-mg group, the last 8 subjects would be enrolled in the third cohort to receive a single 120 mg subcutaneous injection of LY06006.

ELIGIBILITY:
Inclusion Criteria:

* Signed ICF and complied with ICF requirement and restrictions
* Healthy male and female, 18≤age≤65
* In screening visit, male body weight≥50kg，female body weight≥45kg，and 19.0≤BMI≤24.0 kg/m2；
* At screening visit: physical examination, vital signs, laboratory tests, electrocardiogram, chest X-ray examination, abdominal CT examination are normal or abnormal but no clinical significance confirmed by investigators；
* During the study period and within 12 months after the study drug administration, the subjects and partners agreed to use reliable contraceptive measures

Exclusion Criteria:

* Pregnant or lactating women；
* Fertility plan within one year；
* The subject has a history of hypersensitivity or allergy to LY06006 or any of its excipients；or allergy to any drug, food and pollen, or IGE test is positive.
* Subjects are suffering from or have had osteomyelitis or osteonecrosis of the Jaw, or plan to have invasive dental or maxillofacial surgery during the study, or dental or oral surgery wounds unhealed;
* Have fractures in past six months；
* Active respiratory, digestive, urinary, reproductive or skin infections；
* Have oncology family history ；
* Have mental illness history；
* In screening visit: Chest X-ray, abdominal CT indicated clinical significance，for example: tuberculosis, inflammation, et al；
* PPD test positive with 48-72 hrs induration reading≥5mm；
* Blood chemistry：ALT or AST >1.5 ULN，Cr>1.0 ULN；Blood routine：WBC<0.8 LLN or>1.2 ULN；NE<0.8 LLN；PLT<0.8 LLN；HGB<0.8LLN；
* Suffering from or have had the following diseases affecting the bone metabolism: malignant tumors (including myeloma), hypoparathyroidism / hyperthyroidism, hypothyroidism, acromegaly, cushing's syndrome, hypopituitarism, severe chronic obstructive pulmonary disease, rheumatoid arthritis, osteomalacia et al;
* The medicines that may affect bone turnover are used before randomization or planned to use in the study period , including but not limited : denosumab, bisphosphonates or fluorides were used in past 12 months; contraceptives with hormone，hormone replacement therapy（tibolone、hormone、selective estrogen receptor modulators）aromatase inhibitors, calcitonin, strontium salt, parathyroid hormone (or derivative), vitamin D supplement，anabolic steroids, systemic glucocorticoids, calcitriol or analogues, diuretics, anticonvulsant drugs；inhalation or local use of glucocorticoids within 2 weeks
* Significant changes in physical activity in 6 months before randomization; or have been playing strenuous sports, or plan to play strenuous sports during the study period.
* Any of HBsAg, HCV-Ab, Anti-HIV, TP-Ab is positive；
* Hypocalcemia or hypercalcemia，or serum calcium calibrated by serum albumin is not within the normal range
* The average daily smoking amount is more than 5 cigarettes per day during three months before randomization, or smoking can't be prohibited during the study period;
* Alcohol abuse or drank more than 28 units / week of alcohol((1 unit =350ml beer, 45ml spirits or 150ml Wine), or alcohol breath test is positive；
* History of drug dependency or drug abuse, or urine drug screening test is positive；
* Donated whole blood, blood component, or massive hemorrhage （>400ml）three months before randomization.
* Use of any vaccines in 6 months of initiation of study therapy
* participation in another clinical trial within 3 months prior to enrollment
* Had Blood faint and acupuncture syncope history；

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2018-01-10 (Actual); Primary Completion 2019-12-28 (Estimated); Study Completion 2019-12-28 (Estimated)

PRIMARY OUTCOMES:
Number of patients with treatment related adverse events | 56 days
  Number of patients with treatment related adverse events assessed by change from baseline
Number of patients with abnormal laboratory values | 56 days
  Number of patients with abnormal laboratory values assessed by change from baseline

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) | 56 days
Area under the Curve (AUC) | 56 days
Number of patients with anti drug antibodies | 56 days

CONTACTS AND LOCATIONS:
Overall Officials: Huanhuan Jiang, Study Director — Shangdon Boan Biotechnology Co Ltd
Locations (1):
- Peking University People's Hospital, Beijing, Xicheng District, China

IPD SHARING:
Plan to Share IPD: No